CLINICAL TRIAL: NCT05436951
Title: Night Shift Work, On-shift Napping, and Endothelial Function: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Daniel Patterson, PhD, NRP, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY22040156
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Blood Pressure; Endothelial Dysfunction
Keywords: Ambulatory Blood Pressure; Endothelial Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized crossover study design
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-nap, then brief 45-minute nap (Experimental): Participants will be monitored for a total of 48 hours, including a 12-hour simulated night shift. At baseline (consent), participants are randomized to a crossover study design with two study arms (no nap, brief 45-minute nap). In this sequence, participants will perform the 12-hour simulated night shift with no nap first, undergo a minimum of 1-week washout, then return complete the 48-hour protocol again with the brief 45-minute nap.
  Interventions: Behavioral: Brief on-shift nap
- The brief 45-minute nap, then no-nap (Experimental): Participants will be monitored for a total of 48 hours, including a 12-hour simulated night shift. At baseline (consent), participants are randomized to a crossover study design with two study arms (no nap, brief 45-minute nap). In this sequence, participants will perform the 12-hour simulated night shift with the brief 45-minute nap, undergo a 1-week minimum washout, then return to complete the 48-hour protocol again with the no-nap
  Interventions: Behavioral: Brief on-shift nap

INTERVENTIONS:
Behavioral: Brief on-shift nap — The brief nap opportunity will allow for a 45-minute nap between the hours of 0200 and 0300 during the in-lab 12-hour simulated night shift.

SUMMARY:
Cardiovascular disease (CVD) and CVD risk factors such as high blood pressure (BP) are disproportionately higher among night shift workers, including those who work in public safety and healthcare. The purpose of this pilot study is to assess feasibility of collecting data germane to key indicators of cardiovascular health (i.e., ambulatory blood pressure) repeatedly during a simulated night shift protocol. The primary outcome measure will be the number of participants for which at least 70% of required ambulatory BP measures were collected. A result of at least 10 participants/subjects will be considered feasible.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) and CVD risk factors such as high blood pressure (BP) are disproportionately higher among night shift workers, including those who work in public safety and healthcare. Risk of CVD events such as myocardial infarction and stroke are higher among shift workers than non-shift workers. Risk of atrial fibrillation is 1.22 times greater (95%CI 1.02, 1.45) among individuals that work 3-to-8 night shifts per month versus non-shift workers. A comprehensive explanation for why shift workers, especially night shift workers, are at greater risk of CVD is not yet available. However, some research suggests that night shift workers experience repeated exposure to sleep deprivation, which impacts normal patterns in BP and endothelial function. Endothelial dysfunction and disruption of normal BP patterns are independently linked to numerous indicators of CVD, including cardiac-related mortality.

The purpose of this pilot study is to assess feasibility of collecting data germane to key indicators of cardiovascular health (i.e., ambulatory blood pressure) repeatedly during a simulated night shift protocol. Investigators propose a laboratory-based pilot study whereby participants (volunteers) complete two conditions. Condition one will include a 12-hour simulated night shift in our lab with no napping. Condition two will involve a 12-hour simulated night shift in our lab with a 45 minute nap at 0200 hours. Participants will be asked to wear monitoring devices for approximately 48 total hours with the last 12 hours of monitoring (from 1900 to 0700) to be in our lab.

Aim 1: Assess the feasibility of collecting ambulatory BP measures (ABPM) and indicators of endothelial function at multiple time points prior to, during, and after simulated night shift work.

The primary outcome measure will be the number of participants for which at least 70% of required ambulatory BP measures were collected. A result of at least 10 participants/subjects will be considered feasible.

Aim 2: Characterize the impact of simulated night shift work and on-shift napping on BP dipping and endothelial function.

Secondary endpoints include quantifying descriptive statistics (e.g., means and standard deviations) for BP dipping and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

All participants will be working aged adults (18 years of age or older). Investigators are interested in enrolling public safety workers and healthcare workers given how often this group works night shifts.

Criteria that participants will need to address:

1. 18 years of age or older;
2. Currently licensed or certified as an EMS clinician, other public safety shift worker, or other type of healthcare clinicians and actively working in Western Pennsylvania as an EMT, Paramedic, Flight Nurse/Paramedic, other EMS clinician, firefighter, or other type of healthcare clinician (e.g., nurse, physician, physician assistants, patient care technician, or other healthcare clinician);
3. a 'no' answer to #2 above is not a criterion for exclusion.

Exclusion Criteria:

1. Having ever been diagnosed with the following: hypertension, cardiovascular disease, myocardial infarction, stroke/TIA, chronic kidney disease, liver disease, adrenal disease, thyroid disease, rheumatologic disease, hematologic disease, cancer of any type, dementia/memory loss, organ transplantation; major sleep problem; heavy alcohol use; sleep apnea or other diagnosis that is related to problems with breathing or the airway;
2. Current pregnancy;
3. Insomnia is NOT a criterion for exclusion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants for which at least 70% of required Ambulatory BP readings were collected | 48 continuous hours for each arm/condition
  A result of at least 10 participants will be considered feasible

SECONDARY OUTCOMES:
Average blood pressure while awake during simulated night shift | 12 continuous hours for each arm/condition
  The mean and standard deviation of blood pressure measurements taken while participant is awake during the 12-hour simulated night shift
Average blood pressure while napping during simulated night shift | 45 minutes
  The mean and standard deviation of blood pressure measurements taken while participant is napping (sleeping) during the 12-hour simulated night shift that includes the 45-minute nap condition.
Average Reactive Hyperemia Index (RHI) at baseline | 20-30 minutes for each arm/condition
  The mean and standard deviation RHI score for the endothelial dysfunction measurement assessed at baseline
Average Reactive Hyperemia Index (RHI) after simulated night shift | 20-30 minutes for each arm/condition
  The mean and standard deviation RHI score for the endothelial dysfunction measurement assessed after the 12-hour simulated night shift

CONTACTS AND LOCATIONS:
Overall Officials: P. Daniel Patterson, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not have an existing plan to share data after the study has been completed. However, the investigators will develop a process to receive requests for de-identified data from outside investigators once the study has been completed.

REFERENCES:
- [Derived] Patterson PD, Hilditch CJ, Martin SE, Roach DGL, Weaver MD, Okerman TS, Hostler D, Weiss LS, Reis SE. Comparison of 45-min nap versus no-nap during simulated night shift work on endothelial function: a randomized crossover feasibility trial. Pilot Feasibility Stud. 2024 Nov 12;10(1):137. doi: 10.1186/s40814-024-01569-2. PMID 39533414